CLINICAL TRIAL: NCT05595356
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Treatment Resistant Depression: a Randomized Clinical Trial
Brief Title: Home-based Transcranial Direct Current Stimulation for Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210526
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive 30 daily sessions of tDCS. Each session lasts 20 minutes, and delivers a current of 2mA.
  Interventions: Device: transcranial direct current stimulation; Device: run-in sham transcranial direct current stimulation; Behavioral: Psychoeducation video; Behavioral: Tutorial video
- Sham tDCS (Sham Comparator): Participants will receive 30 daily sessions of sham tDCS. Each session lasts 20 minutes, and the sham programming delivers 3 ramps of 30 seconds of active current, the first in the first minute of the session, the second after 10 minutes and the third at the last minute of the session.
  Interventions: Device: sham transcranial direct current stimulation; Device: run-in sham transcranial direct current stimulation; Behavioral: Psychoeducation video; Behavioral: Tutorial video

INTERVENTIONS:
Device: transcranial direct current stimulation — Session description: An electric current of 2mA will be delivered through 35 square centimeters electrodes covered by sponges dampened with saline to reduce impedance. The anode will be placed over the left dorsolateral prefrontal cortex and the cathode will be placed over the right dorsolateral prefrontal cortex. The electrodes will be fixed in a neoprene cap to ascertain their positioning.
  Session duration: 20 minutes
  Frequency of sessions: Daily sessions, from monday to friday, skipping weekends, during 6 weeks.
  Number of sessions: 30 sessions
  The first randomized session will be delivered in the third assessment visit, two weeks after the run-in sham session.
  Other Names: tDCS
  Arms: Active tDCS
Device: sham transcranial direct current stimulation — Session description: Three ramps of 30 seconds of current will be delivered through 35 square centimeters electrodes covered by sponges dampened with saline to reduce impedance. One electrode will be placed over the left dorsolateral prefrontal cortex and the other electrode will be placed over the right dorsolateral prefrontal cortex. The electrodes will be fixed in a neoprene cap to ascertain their positioning.
  Session duration: 20 minutes
  Frequency of sessions: Daily sessions, from monday to friday, skipping weekends, during 6 weeks.
  Number of sessions: 30 sessions
  The first randomized session will be delivered in the third assessment visit, two weeks after the run-in sham session.
  Other Names: sham tDCS, inactive transcranial direct current stimulation
  Arms: Sham tDCS
Device: run-in sham transcranial direct current stimulation — In the second assessment visit, one run-in 20-minute session of sham stimulation, consisting of three ramps of 30 seconds of current, will be delivered through 35 square centimeters electrodes covered by sponges dampened with saline to reduce impedance. One electrode will be placed over the left dorsolateral prefrontal cortex and the other electrode will be placed over the right dorsolateral prefrontal cortex. The electrodes will be fixed in a neoprene cap to ascertain their positioning.
  Other Names: run-in sham tDCS, inactive transcranial direct current stimulation
Behavioral: Psychoeducation video — Watching a video, produced by the research team, containing a brief explanation of what depression is and how it's treated.
Behavioral: Tutorial video — Watching a video, produced by the research team, containing instructions on how to operate de tDCS devices.

SUMMARY:
The aim of this phase II, randomized, double-blind clinical trial is to evaluate the effect of home-based transcranial direct current stimulation (tDCS) in patients with treatment-resistant depression. Major depressive disorder is defined by depressed mood and/or loss of interest in activities, during most of the day, nearly every day, for at least two weeks. It is usually accompanied by other symptoms, such as fatigue, sleep disturbances, thoughts of guilt, suicidal ideation, appetite alterations, difficulty to focus and physical agitation or retardation. It is estimated that its worldwide prevalence is 5%, affecting 280-300 million people. A third of patients with depression will develop treatment resistant depression, where symptoms fail to remit after at least two trials of antidepressants. Beyond psychotropics, another treatment option is neuromodulation, where excitatory or inhibitory signals are delivered to the brain, in order to modulate cortical excitability. The tDCS is a non-invasive brain stimulation method that applies a low intensity direct current (1-2mA) directed to the scalp via the cathode and anode electrodes. The current reaches the cortex, facilitating hyperpolarization or depolarization of the axonal membrane potential. Evidence has shown that this method is presented as a technique able to alter cortical and subcortical neural networks. This technique has been used to treat psychiatric disorders such as depression, bipolar affective disorder, panic, hallucinations, obsessive compulsive disorder, schizophrenia, withdrawal, rehabilitation after stroke and pain syndromes such as neuropathic pain, migraine and fibromyalgia. It has a low cost and less side effects than psychotropic medications. In order to be effective, daily repeated sessions of 20-40 minutes are necessary. When applied in a hospital setting, this frequency of sessions can limit its appliance, especially for depressed patients, whose symptoms include fatigue and loss of interest in activities. Furthermore, transportation costs, frequent absences from work and other activities and overload of the healthcare system would also limit its use. Home based devices are portable and easily operated. Thus, it is possible for patients to administer themselves the treatment, in their own home, everyday. Therefore, the aim of this study is to evaluate the effect of home-based tDCS in treatment resistant depression patients in long-term treatment.

DETAILED DESCRIPTION:
The main outcome is to estimate the variation of the scores of depressive symptoms, measured through the Hamilton Depression Scale with 17 items. Secondary outcomes include response rates, defined as a reduction of at least 50% in scores, and remission rates, defined as a hamilton score lower than 7. Symptom severity, functionality, quality of life and cognitive impairment secondary to depression will also be measured before and after the interventions, as well as inflammatory blood biomarkers and cortical excitability measures. Data from the sessions will be downloaded from the devices to check for treatment adherence.

In the first visit, after being informed by the study and its potential risks, all participants who sign a written informed consent form will undergo a screening interview, to confirm the diagnosis of unipolar major depressive episode and exclude active substance use disorder. A sociodemographic questionnaire will also be applied, for the collection of basic data, clinical comorbidities and use of medications. In the second visit, participants who meet the eligibility requirements will be evaluated for baseline levels of depressive and cognitive symptoms, then undergo one run-in session of sham tDCS (placebo) and receive a wrist actometer that must be used during the following two-week period. After this period, in the third visit, depressive symptoms and actigraphy data will be reassessed, and those who did not wear the wrist actometer for at least 7 consecutive days, and those with an improvement of symptoms superior to 30% will not be included in the rest of the trial due to significant response to one session of placebo. Participants who remain eligible will be randomized in a double blind manner (participant and investigator) in a 1:1 ratio to receive 30 sessions of active tDCS (2mA, for 20 minutes, daily, skipping weekends) or 30 sessions of sham tDCS (inactive current, for 20 minutes, daily, skipping weekends). The first session with the randomized device will be performed under supervision of the study researchers, who will teach the participants how to operate the device, and provide a video with instructions to be watched at home if necessary. A psychoeducation video, produced by the research team, will be sent to all the participants after this visit, containing a brief explanation of what depression is and how it's treated. The aim is to provide information with accessible language and ascertain that all the participants understand their diagnosis, and also understand the role of physical activity, healthy diets and basic sleep hygiene have in the improvement of symptoms. During the next three week period, participants will administer themselves the sessions, from monday to friday. The randomized devices will be programmed to administer daily sessions of 20 minutes, from monday to friday, during 6 weeks. All devices will be programmed to not start sessions on weekends, or run more than one session on the same day, unless stimulation is interrupted by some adversity before it has completed at least 10 minutes. After 10 minutes, even if interrupted abruptly, the session will be considered complete. In order to mimic the side effects of the active stimulation, the sham programming delivers 3 ramps of 30 seconds of active current, the first in the first minute of the session, the second after 10 minutes and the third at the last minute of the session. In the fourth visit, participants return after 3 weeks (15 sessions) of stimulation to reassess symptoms and download device and actigraphy data. Participants will return to their homes to administer the following 15 sessions and return after three weeks for the fifth visit, when depressive and cognitive symptoms will be reassessed and participants will be asked if they believe they receive active or sham stimulation. The sixth and last visit takes place 3 months after the end of the trial, for follow up on symptoms and another 15 days of actigraphy for monitoring sleep patterns. Between the third and the fifth visits, weekly online questionnaires will be sent to the participants, for the evaluation and monitoring of adverse effects during the trial. Blood samples and cortical excitability measures (assessed through TMS) will be collected twice, in the third and fifth visits (before and after the trial). During the whole trial, online support via whatsapp will be provided. Members of the team will be available for answering questions and doubts that should arise anytime during the treatment. During the trial, no alterations will be made to the participants' prescriptions, to prevent response to medication as a confounding factor. Participants presenting acute risk or worsening of symptoms at any time point will be removed from the study and receive standard care measures by the research team.

All the questionnaires and patient sensitive data will be collected through the REDCap platform. Anonymous data regarding the adherence to treatment sessions will be stored in an institutional Google Drive cloud. For the statistical analysis, the database will be downloaded with anonymized data. R software and SPSS version 21 will be used. Analyses will be performed considering intention to treat and last observation carried forward will be used in cases of missing data. Distribution of variables will be described in means, medians, standard deviations, interquartile ranges, frequencies and proportions, as appropriate. Multilevel Mixed-Effects Linear Regression or Generalized Estimating Equations will be used to evaluate the time*group interactions for depressive symptoms. Secondary outcomes will be evaluated through multiple linear regressions. Bonferroni test for multiple comparisons will be used to detect differences between groups in all timepoints.The level of statistical significance was established as p < 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Current diagnosis of Major Depressive Episode according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) criteria
* Presence of depressive symptoms that did not improve after at least two trials of first line antidepressants, for at least four weeks each, in optimized doses
* Patients living in Porto Alegre or its metropolitan region
* No changes in prescription in the last four weeks upon entering the trial

Exclusion Criteria:

* Psychotic symptoms
* Acute risk, or indication of hospitalization
* Diagnosis of current Substance Use Disorder (alcohol, marijuana, cocaine, sedatives/hypnotics, stimulants, inhalants and others) according to DSM-V criteria
* Presence of metallic implants or medical devices implanted in the brain
* Pacemakers and cochlear implants
* Neurological diseases: epilepsy, malformations
* History of head trauma or neurosurgery
* Pregnancy
* Cognitive impairment severe enough to prevent the operation of the tDCS device without professional assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in scores obtained in the Hamilton Depression Rating Scale | Assessed in visit 2 (baseline pre-sham stimulation, week 0), visit 3 (baseline post-sham stimulation, week 2), visit 4 (middle of the trial, week 5), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in depressive symptoms, measured by the 17-item version of the Hamilton Depression Rating Scale, before, during and after application of home-based tDCS. The score values ranges from 0 to 49, and higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Change in scores in the Patient Health Questionnaire - 9 | Assessed in visit 2 (baseline pre-sham stimulation, week 0), visit 3 (baseline post-sham stimulation, week 2), visit 4 (middle of the trial, week 5), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in depressive symptoms, measured by the Patient Health Questionnaire 9-item, before, during and after application of home-based tDCS. The score values ranges from 0 to 30, and higher scores represent worse outcomes.
Change in Clinical Global Impression of Severity scores | Assessed in visit 2 (baseline pre-sham stimulation, week 0), visit 4 (middle of the trial, week 5), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in severity of clinical depression symptoms, before, during and after application of home-based tDCS. The score values ranges from 1 to 7, and higher scores represent worse outcomes.
Change in the Eurohis-Quality of Life Index | Assessed in visit 2 (baseline pre-sham stimulation, week 0), visit 4 (middle of the trial, week 5) and visit 5 (upon trial completion, week 8)
  Change in quality of life perception measured by the Eurohis-Quality of Life Index, a 8-item questionnaire, before and after application of home-based tDCS. The score values ranges from 8 to 40, and higher scores represent better outcomes.
Change in the 12-item World Health Organization Disability Assessment Schedule II | Assessed in visit 2 (baseline pre-sham stimulation, week 0), visit 4 (middle of the trial, week 5) and visit 5 (upon trial completion, week 8)
  Change in disability scores measured through the 12 item World Health Organization Disability Assessment Schedule II, before, during and after application of home-based tDCS. The score values ranges from 12 to 60, and higher scores represent worse outcomes.
Change in the Screen for Cognitive Impairment in Psychiatry | Assessed in visit 2 (baseline pre-sham stimulation, week 0) and visit 5 (upon trial completion, week 8)
  Change in cognitive symptoms measured through the Screen for Cognitive Impairment in Psychiatry, before and after application of home-based tDCS. The answers are converted into Z-Scores, and higher scores represent better outcomes.
Change in the Mood Rhythm Instrument | Assessed in visit 3 (baseline post-sham stimulation, week 2), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in mood and behaviour rhythms measured through the Mood Rhythm Instrument, before and after application of home-based tDCS.
Change in the Ultra-short Munich ChronoType Questionnaire | Assessed in visit 3 (baseline post-sham stimulation, week 2), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Changes in periods of activity and rest, measured through the Ultra-short Munich ChronoType Questionnaire, before and after application of home-based tDCS. This questionnaire records the sleep and wake times of the participants, to calculate the total sleep time and variations in the circadian cycle.
Change in the Sleep Hygiene Index | Assessed in visit 3 (baseline post-sham stimulation, week 2), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in sleep related behaviours, measured through the Sleep Hygiene Index, before and after application of home-based tDCS. The score values ranges from 13 to 65, and higher scores represent worse outcomes.
Change in Insomnia Severity Index | Assessed in visit 3 (baseline post-sham stimulation, week 2), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in insomnia symptoms measured through the Insomnia Severity Index, before and after application of home-based tDCS. The score values ranges from 0 to 28, and higher scores represent worse outcomes.
Change in quality of sleep | Assessed in visit 3 (baseline post-sham stimulation, week 2), visit 5 (upon trial completion, week 8) and visit 6 (3 months after trial completion)
  Change in quality of sleep, measured through the Sleep Quality component of the Pittsburgh Sleep Quality Index, before and after application of home-based tDCS. The score values ranges from 1 to 4, and higher scores represent worse outcomes.
Actigraphy measures | Continuous monitoring during the 8 weeks from visit 2 through visit 5, and during the 2 weeks before visit 6
  Changes in periods of activity and rest, monitored by portable actigraphy devices, before and after application of home-based tDCS
Changes in cortical excitability: motor threshold | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Changes in motor threshold (a cortical excitability measure) assessed through magnetic transcranial stimulation, before and after application of home-based tDCS.
Changes in cortical excitability: silent period | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Changes in silent period (a cortical excitability measure) assessed through magnetic transcranial stimulation, before and after application of home-based tDCS.
Changes in cortical excitability: motor evoked potential | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Changes in motor evoked potential (a cortical excitability measure) assessed through magnetic transcranial stimulation, before and after application of home-based tDCS.
Serum levels of Brain Derived Neurotrophic Factor (BDNF) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of BDNF before and after application of home-based tDCS
Serum levels of calcium-binding protein B (S100B) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of S100B before and after application of home-based tDCS
Serum levels of Interleukine 1-beta (IL-1b) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of IL-1b before and after application of home-based tDCS
Serum levels of Interleukine 6 (IL-6) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of IL-6 before and after application of home-based tDCS
Serum levels of Tumor Necrosis Factor (TNF-α) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of TNF-α before and after application of home-based tDCS
Serum levels of C-reactive protein (CRP) | Assessed in visit 3 (baseline post-sham stimulation, week 2) and visit 5 (upon trial completion, week 8)
  Measurement of serum levels of CRP before and after application of home-based tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Pio de Almeida Fleck, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No